CLINICAL TRIAL: NCT04228393
Title: The Individualized Treatment of 6-mercaptopurine in Children With Acute Lymphoblastic Leukemia in China
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wei Zhao (Other)
Collaborators: Institute of Hematology & Blood Diseases Hospital, China (Other); Qianfoshan Hospital (Other); Qilu Hospital of Shandong University (Other); Children's Hospital of Hebei Province (Other); The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor-Investigator, Wei Zhao, Professor; Head of department of clinical pharmacy and pharmacology, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-6-mercaptopurine-001
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
Keywords: acute lymphoblastic leukemia; 6-mercaptopurine; children; individualized treatment
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment regimen (Active Comparator): 6-mercaptopurine was administered according to the Chinese Children Cancer Group (CCCG) protocol-ALL 2015.
  Interventions: Drug: 6-mercaptopurine; Procedure: Standard treatment
- Individualized treatment regimen (Experimental): 6-mercaptopurine was administered on the basis of Chinese Children Cancer Group (CCCG) protocol-ALL 2015 combined with Clinical Pharmacogenetics Implementation Consortium (CPIC), genotypes and the concentrations of 6-TGN in red blood cells.
  Interventions: Drug: 6-mercaptopurine; Procedure: Individualized treatment

INTERVENTIONS:
Drug: 6-mercaptopurine — 6-mercaptopurine was administered orally to patients once daily.
  Other Names: 6-MP
Procedure: Standard treatment — The initial dose is 50mg/m2. The dose was adjusted according to white blood cells.
  Arms: Standard treatment regimen
Procedure: Individualized treatment — The initial dose is determined according to the genotypes of patients combined with Clinical Pharmacogenetics Implementation Consortium (CPIC). The dose was adjusted according to white blood cells, genotypes and the concentrations of 6-TGN in red blood cells.
  Arms: Individualized treatment regimen

SUMMARY:
The purpose of this study was to assess the efficacy and safety of individualized treatment of 6-mercaptopurine (6-MP) in Chinese children with acute lymphoblastic leukemia, and to investigate the dose-concentration-response (DER) relationship between thiopurine metabolites and adverse events. The individualized administration of 6-MP was established in Chinese children with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
To inflict minimal pain on the child contributing blood samples, opportunistic sampling design was chosen to collect pharmacokinetic samples.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of acute lymphoblastic leukemia;
2. Age 1-18y at time of initial diagnosis;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
4. Informed consent signed by the patients parents or guardians before initiation of the study.

Exclusion Criteria:

1. Ph-positive ALL, matrue B-cell ALL, BC-CML;
2. Secondary to immunodeficiency, second cancer；
3. Abnormal liver and kidney function;
4. Patients divided into intermediate or high risk groups according to the risk grouping criteria of the Chinese Children Cancer Group (CCCG) protocol-ALL 2015;
5. Patients who enrolled in another clinical trial;
6. Expected survival time less than the treatment cycle;
7. Patients with other factors that researcher considers unsuitable for inclusion

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
leukopenia | 6 weeks
  Leukopenia was graded by common toxicity criteria as follows: Grade 3, 1.0-2.0 × 109/L, and Grade 4, < 1.0 × 109/L.
thiopurine-induced leukopenia | 6-weeks
  Resolution of leukopenia was determined after 6-MP dose reduction or discontinuation, both in the absence of other apparent causes for the leukopenia or its disappearance.

SECONDARY OUTCOMES:
hepatotoxicity | 6 weeks
  Hepatotoxicity was defined as aspartate aminotransferase (AST) or alanine transaminase (ALT) levels 2-fold above the upper limit without cytolysis.
6-thioguanine nucleotides (6-TGN) concentrations in erythrocytes. | 3 months
  Peripheral blood samples were obtained from steady-state plasma concentrates by opportunistic sampling design.
6-methylmercaptopurine nucleotides (6-MMPN) concentrations in erythrocytes. | 3 months
  Peripheral blood samples were obtained from steady-state plasma concentrates by opportunistic sampling design.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Ph.D, Principal Investigator — Shandong University
Locations (1):
- State Key Laboratory of Experimental Haematology, Department of Paediatric Haematology, Institute of Haematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tanjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Zhou Y, Wang L, Sun LR, Zhang L, Wang HM, Liu XT, Yang F, Wu KL, Liang YL, Zhao BB, Zhuang Y, Fu JQ, Song C, Li Y, Wang LZ, Xu HJ, Gu Y, van den Anker J, Ju XL, Zhu XF, Zhao W. Individualized Use of 6-Mercaptopurine in Chinese Children with ALL: A Multicenter Randomized Controlled Trial. Clin Pharmacol Ther. 2024 Feb;115(2):213-220. doi: 10.1002/cpt.3061. Epub 2023 Oct 16. PMID 37753808